CLINICAL TRIAL: NCT01445886
Title: Evaluation of the Efficacy and Safety of Indigo Naturalis Oil Extract and Calcipotriol Solution in Patients With Nail Psoriasis
Brief Title: Comparison of Indigo Naturalis Oil Extract and Calcipotriol Solution in Treating Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yin-ku Lin (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Sponsor-Investigator, Yin-ku Lin, Chief of Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG2A0191
Record Dates: First submitted 2011-04-25; First posted 2011-10-04 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Nail Psoriasis
Keywords: Nail Psoriasis; Indigo Naturalis; Indirubin; Calcipotriol; Nail Psoriasis Severity Index
MeSH Terms: interventions — Oils; calcipotriene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indigo Naturalis Extract in Oil (Experimental): A 5-ml eye drop bottles contain indigo naturalis powder mixed with olive oil, and the concentration was 200 ug indirubin per ml. Each subject was asked to apply one to two drops (0.05 ml per drop) of the solution twice daily onto the nail folds, plus the hyponychium, of affected nails. The maximum period of treatment was 24 weeks or until there was complete clearing of their nail psoriasis.
  Interventions: Drug: Indigo Naturalis Extract in Oil
- Calcipotriol solution (Active Comparator): Calcipotriol solution (Daivonex® scalp solution, calcipotriol 50 ug/ml) was purchased from LEO Pharmaceutical Products, Ltd. (Ballerupt, Denmark) and also distributed into 5-ml eye drop bottles for this trial.Each subject was asked to apply one to two drops (0.05 ml per drop) of the solution twice daily onto the nail folds, plus the hyponychium, of affected nails. The maximum period of treatment was 24 weeks or until there was complete clearing of their nail psoriasis.
  Interventions: Drug: Calcipotriol Solution

INTERVENTIONS:
Drug: Indigo Naturalis Extract in Oil — The participants applied indigo naturalis extract in oil topically to one of two bilaterally symmetrical psoriatic finger nails twice daily for 24 weeks.
  Other Names: Lindioil
  Arms: Indigo Naturalis Extract in Oil
Drug: Calcipotriol Solution — The participants applied calcipotriol solution topically to one of two bilaterally symmetrical psoriatic finger nails twice daily for 24 weeks.
  Other Names: Calcipotriol
  Arms: Calcipotriol solution

SUMMARY:
The purpose of this study is to compare the efficacy and safety of indigo naturalis oil extract and calcipotriol solution in the treatment of psoriatic nails, to show that indigo naturalis oil extract may be a good choice for treating nail psoriasis, and potentially an effective alternative for those who do not respond well to traditional therapy.

DETAILED DESCRIPTION:
In the literature, the efficacy of traditional Chinese medicine in treating nail psoriasis is rarely reported. Recently, the investigators developed a new product, indigo naturalis oil extract, which worked well in nail disease. In our randomized, observer-blind, vehicle-controlled trial showed that indigo naturalis oil extract is effective and safe in treating nail psoriasis. This study aims to compare the efficacy and safety of indigo naturalis oil extract with calcipotriol solution in patients with nail psoriasis using controlled, bilateral comparison

The investigators will enroll 33 patients with nail psoriasis from the ambulatory department of Chang Gung Memorial Hospital. Indigo naturalis oil extract will be consistently applied on either the left or right affected nail folds, while calcipotriol will be applied on the opposite side, both twice daily for 24 weeks, allowing intra-patient comparison. The nails will be assessed by two dermatologists before treatment and at week 2, 4, 8, 12, 16, 20, 24.

ELIGIBILITY:
Inclusion Criteria:

1. Nail psoriasis of the matrix and/or of the nail bed in at least one fingernail.
2. Good general health.
3. Agreement to avoid pregnancy for the study duration

Exclusion Criteria:

1. Concomitant topical treatment (corticosteroids), phototherapy, or any systemic treatment (retinoids, cyclosporine, methotrexate, systemic corticosteroids and biological agents) that could affect nail psoriasis.
2. Patients with severe hepatic or renal disorders.
3. Lactating, pregnant or planning pregnancy
4. Unwillingness to comply with study protocol.
5. A history of sensitivity to indigo naturalis. -

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ku Lin, M.D., Ph.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Derived] Lin YK, Chang YC, Hui RC, See LC, Chang CJ, Yang CH, Huang YH. A Chinese Herb, Indigo Naturalis, Extracted in Oil (Lindioil) Used Topically to Treat Psoriatic Nails: A Randomized Clinical Trial. JAMA Dermatol. 2015 Jun;151(6):672-4. doi: 10.1001/jamadermatol.2014.5460. No abstract available. PMID 25738921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with nail psoriasis were recruited from the outpatient Department of Traditional Chinese Medicine and Dermatology at the Chang Gung Memorial Hospital (CGMH), Taiwan from January 2011 to May 2012.
Pre-assignment Details: This study screened 43 subjects with 33 recruited, and 28 subjects finished the study. ( 2 failure to return, 7 violation of selection criteria at entry, 3 other protocol violation and 3 refused treatment/withdraw violation)
Groups:
- Indigo Naturalis Extract in Oil VS Calcipotriol: Patients were instructed to apply Lindioil (indigo naturalis extract in oil) to the fingernails of one hand (experimental group) and calcipotriol solution to the fingernails of the other hand (control group) twice daily for 24 weeks.
Period: Overall Study
Arm/Group | Indigo Naturalis Extract in Oil VS Calcipotriol
Started | 33
Completed | 28
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Indigo Naturalis Extract in Oil VS Calcipotriol
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Single-handed Nail Psoriasis Severity Index (shNAPSI) at 24 Weeks
Description: The nails will be assessed by two dermatologists at baseline and after treatment 4, 8, 12, 16, 20, 24 weeks using single-handed Nail Psoriasis Severity Index (shNAPSI) score. shNAPSI evaluation: Each nail is given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) , the total of which is the score for that nail (0-8); the range of shNAPSI of one hand is between 0 and 40, with higher score indicating more severe symptoms. Nail bed psoriasis: presence of any of the nail bed features (onycholysis, hemorrhages, hyperkeratosis, "oil drop" (salmon patch dyschroma): 0 for none, 1 for 1 quadrant only, 2 for 2 quadrants, 3 for 3 quadrants, and 4 for 4 quadrants. Nail matrix psoriasis: presence of any of the nail matrix features (pitting, leukonychia red spots in the lunula, crumbling): 0 for none, 1 if present in 1 quadrant of the nail, 2 if present in 2 quadrants of the nail, 3 if present in 3 quadrants of the nail, and 4 if present in 4 quadrants of the nail.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Indigo Naturalis Oil Extract: Indigo Naturalis Oil Extract: The participants applied indigo naturalis oil extract topically to one of two bilaterally symmetrical psoriatic finger nails twice daily for 24 weeks.
Arm/Group | Indigo Naturalis Oil Extract | Calcipotriol Solution
Number analyzed (Participants) | 33 | 33
units on a scale
  baseline | 27.2 (7.83) | 27.4 (8.55)
  week 24 | 14.4 (8.85) | 20.4 (8.47)

2. Secondary Outcome: Change From Baseline in Modified Target NAPSI for the Single Most Severely Affected Nail
Description: The target nail will be assessed by two dermatologists before treatment and at week 4, 8, 12, 16, 20, 24 using modified target NAPSI score (mtNAPSI, 0-96).
  mtNAPSI evaluation: a target nail is divided into 4 quadrants and for each quadrant the nail parameters (oil drop, onycholysis, hyperkeratosis, hemorrhages, pitting, leukonychia, red spots on the lunula, and crumbling) are assessed separately: 0 = no sign, 1 = mild, 2 = moderate, and 3 = severe; the range of mtNAPSI is between 0 and 96, with higher score indicating more severe symptoms.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Indigo Naturalis Oil Extract | Calcipotriol Solution
Number analyzed (Participants) | 33 | 33
units on a scale
  baseline | 17.7 (6.17) | 16.9 (6.45)
  week 24 | 5.9 (4.11) | 9.5 (5.16)

3. Secondary Outcome: Physician's and Subject's Global Assessment
Description: The Physician's and Subject's Global Assessment (PGA and SGA) will be assessed by two dermatologists and participant himself/herself respectively after treatment 24 weeks.
  A 6-point scale was used for both SGA and PGA: 0 = worse, 1 = 0-24% clearing with little or no change, 2 = 25-49% clearing with slight improvement, 3 = 50-74% clearing with moderate improvement, 4 = 75-99% clearing with striking improvement, 5 = cleared. A score between 3 and 5 was considered to be a positive response and a score between 0 and 2 a poor response.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Indigo Naturalis Oil Extract | Calcipotriol Solution
Number analyzed (Participants) | 28 | 28
units on a scale
  PGA 1 | 3.7 (0.82) | 2.5 (1.26)
  PGA 2 | 3.4 (1.10) | 2.3 (1.36)
  SGA | 3.9 (0.76) | 2.6 (1.23)

ADVERSE EVENTS:
Time Frame: Baseline and Week 24
Arm/Group | Indigo Naturalis Oil Extract | Calcipotriol Solution
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes